#### 1. Protocol details

#### PROTOCOL TITLE: 1.1

Personalised simulation technologies for optimising treatment in the inte

# 1.2 Names (titles), roles and contact details of:

#### **Sponsor**

Guy's and St Thomas' NHS Foundation Trust

Elizabeth Bruna 16th floor Tower Wing Guy's Hospital Great Maze Pond London SE1 9RT

## r&d@gstt.nhs.uk

02071887188

#### **Chief Investigator**

Dr Luigi Camporota

Intensive Care Research Office Ground Floor South Wing Block C, Lane Fox Unit, St Thomas' Hospital, Westminster Bridge Road, London, **United Kingdom** SE1 7EH

luigi.camporota@gstt.nhs.uk 020 7188 3046

N

## 1.3 Protocol details

Version number 1.0

Draft

Date 05/02/2020

#### N

# 2 Signature Page

The Chief Investigator and the R&D (sponsor office) have discussed this agree to perform the investigations and to abide by this protocol

The investigator agrees to conduct the trial in compliance with the approx Data Protection Act (1998), the Trust Information Governance Policy (or Research Governance Framework (2005' 2<sup>nd</sup> Edition; as amended), the regulatory requirements as amended.

| Chief investigator | |
|------------------------|-----------|
| Dr Luigi Camporota | |
| | Signature |
| Sponsor Representative | |
| R&D to Add | |
| GSTFT | Signature |

# **Contents Page**

9.1

| 1. Pro | tocol details |
|---------|-----------------------------------------------|
| 1.1 | PROTOCOL TITLE: |
| 1.2 | Names (titles), roles and contact details of: |
| 1.3 | Protocol details |
| 2 Sign | nature Page |
| Content | s Page |
| 3 List | of Abbreviations and Definitions |
| 4 Sur | nmary/Synopsis |
| 5 Inti | roduction |
| 6 Stu | dy objectives and purpose |
| 7 Stu | dy design & Flowchart |
| 7.1 | Study Design |
| 7.2 | Flowchart |
| 8 Suk | pject selection |
| 8.1 | Inclusion Criteria |
| 8.2 | Exclusion Criteria |
| 9 Stu | dy procedures |

Subject recruitment and screening.....

| 11.1.3 | Ventilator |
|----------|-----------------------------------------------|
| 11.1.4 | Blood Gas Analysis |
| 11.1.1 | ECMO |
| 11.2 For | mat and Scale of Data |
| 11.3 Me | thodologies of Data Collection and Generation |
| 11.4 Dat | ta Quality and Standards |
| 11.5 Dat | ta handling and record keeping |
| 11.5.1 | GSTFT |
| 11.5.2 | Data Repository |
| 11.5.3 | Academic Partners |
| 11.6 Me | tadata standards and data documentation |
| 11.6.1 | Data Set Directory Structures and Filenames |
| 11.6.2 | Metadata Descriptive Files |
| 11.7 Dat | ta preservation strategy and standards |
| 11.7.1 | GSTFT |
| 11.7.2 | Data Repository |
| 11.7.3 | Academic Collaborators |

Demographics .....

Physiological .....

11.1.1

11.1.2

| | п |
|---|---|
| n | ı |
| m | м |

| 14 | Financing and Insurance |
|------------|-----------------------------|
| 15 | Reporting and dissemination |
| References | |

# 3 List of Abbreviations and Definitions

GSTFT Guy's and St Thomas' NHS Foundation Trust

UON University of Nottingham

UWAR University of Warwick

# 4 Summary/Synopsis

| Title | Personalised simulation technology |
|------------------------------------|------------------------------------|
| | intensive care unit |
| Protocol Short Title/Acronym | PSTOTICU |
| Protocol Version number and Date | 0.1.4 21/08/2019 |
| IRAS Number | 266780 |
| REC Reference | NA |
| Study Duration | 2 years |
| Sponsor name | Guy's and St Thomas' NHS Foun |
| Chief Investigator | Dr Luigi Camporota |
| Funder | Engineering and Physical Science |
| Medical condition or disease under | Respiratory Failure |
| investigation | |
| Purpose of research | This study aims to further dev |
| | models, by the fitting of those m |
| | data of critical care patients. |
| Primary objective | To further develop our simulation |
| | of recently proposed therapeuti |
| Secondary objective (s) | To integrate data-streams and c |
| | our existing modelling technology |
| | individual patients and treatme |
| | imminent problems. |
| | To develop mathematical me |
| | explore the "design space" of p |
| | individual patient in simulation, |
| | can be suggested for evaluation |
| Number of Episodes | 5,000 |
| Study Type | Observational |
| Endpoints | Not Applicable |
| Main Inclusion Criteria | This project will include crit |

#### 5 Introduction

This project aims to further develop and refine in silico physiological moment models to the physiological and treatment data of critical care patients. development is fitting the model to, and its description of, the physiological interventions. An example would be how a patients physiological increase in positive end expiratory pressure (PEEP). Data for this exphysiological and treatment data pre and post ventilator changes (e.g., PE the clinical team, for a clinically appropriate time period.

Computer simulation offers a new approach to traditional medical rese suited to investigating treatment of critical illness. Critically ill patients great detail, providing extensive, high quality data streams for model patient-matching. Models based on this data can incorporate very compl be validated against responses of individual patients, for use as investiga

In contrast to trials on animal models and humans, in silico models of disease pathology are completely configurable, reproducible and reusable combinations of treatments, can be applied to the same patient or subset to understand mode of action, quantitatively compare effectiveness in variative variations for particular clinical objectives and particular patient grounds.

It is widely accepted that modification of existing mechanical ventilation novel physical treatment strategies could significantly reduce pulmo impairment, and mortality rates, particularly if combined with novel pha-

To achieve this we are undertaking a collaborative project between three different and complimentary areas of expertise.

The three institutions involved in this project are:

# 6 Study objectives and purpose

This project is a collaborative endeavour between Guy's and St Thomas academic collaborators at the University of Nottingham and the University further develop and refine in silico physiological models, by the fitti physiological and treatment data of critical care patients.

The project's primary objective is to further develop our simulation simulation of commonly used therapeutic interventions within the in amenable interventions include prone positioning, optimising the cobreathing effort with mechanical ventilation, application of recruitment cause and maintain an "open lung", and Extra-corporeal membrane interventions have been chosen on the basis of amenability to an optimisation, possessing a strong potential for providing improvement in current usage in many ICU's worldwide.

real time simulation of individual patients and treatments. Sufficient models would enable systematic and efficient exploration of the possible for an individual patient in simulation, allowing optimised treatment streadly evaluation by the clinician. Possible therapeutic interventions to be explosed pulmonary recruitment (alveolar re-opening) manoeuvres, venue, a airway-pressure release ventilation low tidal volume, high positi

Integration of available data within the ICU with our existing modelling t

inspiratory flow waveform modification, and closed-loop ventilatory con-To facilitate the further development of the simulation platform requires

curated data sets representative of the therapeutic interventions of interventions of interventions of interventions of interventions of interventions are collated to catalogue and share collated data sets between corepository will enforce the oversight and governance ensuring the requence protection against unlawful or unauthorised processing, access, loss, des

At this stage of the project, the simulation platform will not be accessib

# 7 Study design & Flowchart

## 7.1 Study Design

This study aims to further develop and refine in silico physiological mo models to the physiological and treatment data of critical care patients.

Of specific interest to model development is fitting the model to, physiological response of patients to specific interventions. An exampl physiological parameters respond to an increase in PEEP. Data for this e physiological and treatment data pre and post ventilator changes (e.g., PE the clinical team, for a clinically appropriate time period. This would com

Data required for this study will therefore be truncated case report data short time periods, on the order of 12 hours duration. The exact lengtl determined by the clinical scenario, but would be for a clinically appropr

No attempt will be made to capture data from entire patient cohorts or t

There is no intention to implement any study specific interventions or tre be retrospective, pragmatic and limited to that data recorded throu routinely provided to all patients.

Within this project, there is no intention for physiological models develop Clinicians will have no access or exposure to the simulations and predicti by the models that this project aims to develop.

For the purposes of this document, a data set is defined as a collated se subject and one intervention.

#### 7.2 Flowchart

The collaborative nature of this study requires that data be managed a environments:

N



# 8 Subject selection

Subjects will be drawn from the adult critical care population at GSTFT. S receiving mechanical ventilation.

It is anticipated that this project will require several iterations of development, with each iteration examining a different treatment intervial will inform the exact nature of data collection in the subsequent iteration and analysis iterations that will be required is dependent on the development.

As noted in section 7.1 collated data sets will episodic in nature with exthe order of twelve hours. It is entirely possible that the admission and diseveral episodes of interest, or the patient may receive a similar interver episodes may be therefore be contributed under differing study ids to catalogued in the data repository.

#### 8.1 Inclusion Criteria

- At least 18 years of age
- Patients admitted to GSTFT Intensive Care between th 31/03/2019
- · Receiving mechanical ventilation

#### 8.2 Exclusion Criteria

Pregnancy or lactation.

# 9 Study procedures

## 9.1 Subject recruitment and screening

Episodes of interest will be identified retrospectively by querying existing attributes. As an example, patient treatment data could be queried for episetting is increased from 5 to 10.

Data subjects will not be approached as data is collected retrospectively existing data sources. We will not be requested any additional data or re

Consent will not be sought from individual patients due to the non-inte nature of the data collection.

Data collection will be limited to that data recorded as part of routi 01/01/2010 and 31/03/2019

## 9.2 Schedule of assessments for each visit

Data is available from the electronic health records and the data export technology employed in the routine care of critically ill patients.

No schedule of assessment is planned due to the retrospective nature of health care records.

# 9.3 Follow up Procedures

There are no follow up procedures planned for this study.

# 9.4 End of Study Definition

Completion of the project is defined as the time point five years after cactivities.

# 10 Assessment of Safety

Study procedures for this study consist of data collection from the electron in the routine care provided to patients. It is anticipated that this study patient safety than that caused by their routine clinical care.

## 10.1 Study Steering Committee

There will be no monitoring, steering or safety committees set up for this

# 10.2 Ethics & Regulatory Approvals

Appropriate HRA and REC will be in place before the study commences.

#### 11 Data

#### 11.1 Data to be collected

Data will be collected within four domains:

- Demographics
- Physiological
- Ventilation
- Blood gas analysis

Demographic data will be collected from the health care record, and is of

Physiological data is continuously captured by monitoring equipment (Phi within ICU, and recorded on a regular basis into an electronic health red Data can also be captured remotely from the continuous stream capture

Ventilator parameters and patient ventilatory parameters are measured at the bedside in the ICU by the patient ventilators (Drager V500). This c basis into an electronic health record system by clinical staff. Data can from the ventilators.

Blood gas analysis results are collected routinely as part of the care of ICU their electronic health record. Data will be collected retrospectively from

Data points that will be collected from each domain are detailed below. identify specific data fields, alongside a short description of that data realistic that only subsets of the entire list of potential data fields will

present in individual data sets, with availability dependent on differing page 1

#### 11.1.1 Demographics

Invasive mean blood pressure m

Invasive systolic blood pressure

| CENTRAL_TEMP_MONITOR_C | Central temperature measureme |
|---------------------------|------------------------------------|
| PERIPHERAL_TEMP_MONITOR_C | Peripheral temperature measure |
| ECG_HEART_RATE_MIN | ECG Heart Rate |
| HEART_RATE_MONITOR_MIN | Monitor Heart Rate |
| ECG_RHYTHM_MONITOR | ECG cardiac rhythm |
| PVC_RATE_MONITOR_MIN | Premature Ventricular Contraction |
| ECTOPIC_BEAT_MONITOR_STR | Premature Ventricular Contraction |
| ECT_RATE_MONITOR_MIN | ECG Ectopic Rate |
| SPO2_MONITOR monitoring | Photoplethysmogram - Non-ii |
| RESP_RATE_MONITOR_MIN | Respiratory Rate |
| NIBP_SYS_MMHG | Non-invasive systolic blood press |
| NIBP_DIA_MMHG | Non-invasive diastolic blood pres |
| NIBP_MEAN_MMHG | Non-invasive mean blood pressu |
| ABP_SYS_MMHG | Invasive systolic blood pressure i |
| ABP_DIA_MMHG | Invasive diastolic blood pressure |

ART\_DIA\_MMHG Invasive diastolic blood pressure ART\_MEAN\_MMHG Invasive mean blood pressure m

ABP\_MEAN\_MMHG

ART\_SYS\_MMHG

| CENTRAL_TEMP_ICIP_C | Central temperature measureme |
|------------------------|------------------------------------|
| PERIPHERAL_TEMP_ICIP_C | Peripheral temperature measure |
| HEART_RATE_ICIP | Heart Rate |
| CARDIAC_RHYTHM_ICIP | Cardiac Rhythm |
| SPO2_ICIP | Photoplethysmogram |
| NIBP_SYS_ICIP_MMHG | Non-invasive systolic blood press |
| NIBP_DIA_ICIP_MMHG | Non-invasive diastolic blood pres |
| NIBP_MEAN_ICIP_MMHG | Non-invasive mean blood pressu |
| ABP_SYS_ICIP_MMHG | Invasive systolic blood pressure i |
| ABP_DIA_ICIP_MMHG | Invasive diastolic blood pressure |
| ABP_MEAN_ICIP_MMHG | Invasive mean blood pressure m |
| ART_SYS_ICIP_MMHG | Invasive systolic blood pressure i |
| ART_DIA_ICIP_MMHG | Invasive diastolic blood pressure |
| ART_MEAN_ICIP_MMHG | Invasive mean blood pressure m |

PABP\_SYS\_ICIP\_MMHG Systolic pulmonary artery blood PABP\_DIA\_ICIP\_MMHG Diastolic pulmonary artery blood Mean pulmonary artery blood p PABP\_MEAN\_ICIP\_MMHG

CVP\_MEAN\_ICIP\_MMHG Invasive central venous pressure

CARDIAC\_OUTPUT\_ICIP\_L\_MIN Cardiac Output

**Pressure Low** 

Pressure High

Pressure mean

| P_MIN_CMH2O | Pressure minimum |
|----------------------------|---------------------------------|
| P_PEAK_CMH2O | Pressure peak inspiratory |
| P_PLATEAU_CMH2O | Pressure plateau |
| MIN_VOL_EXP_L_MIN | Expired minute volume |
| MIN_VOL_EXP_SPON_L_MIN | Expired minute volume - sponta |
| MIN_VOL_EXP_MAND_L_MIN | Expired minute volume - manda |
| MIN_VOL_LEAK_L_MIN | Minute volume leak |
| TIDAL_VOLUME_MLS | Tidal Volume |
| TIDAL_VOLUME_INSP_MLS | Tidal Volume Inspired |
| TIDAL_VOLUME_EXP_MLS | Tidal Volume Expired |
| TIDAL_VOLUME_SPON_MLS | Tidal Volume Spontaneous |
| TIDAL_VOLUME_INSP_SPON_MLS | Tidal Volume Inspired Spontaneo |
| TIDAL_VOLUME_EXP_SPON_MLS | Tidal Volume Expired Spontaneo |
| TIDAL_VOLUME_MAND_MLS | Tidal Volume Mandatory |
| TIDAL_VOLUME_INSP_MAND_MLS | Tidal Volume Inspired Mandator |
| TIDAL_VOLUME_EXP_MAND_MLS | Tidal Volume Expired Mandatory |

P\_LOW\_CMH2O

P\_HIGH\_CMH2O

P\_MEAN\_CMH2O

| E_IE | Expiratory component IE ratio |
|--------------------|--------------------------------|
| I_IE_SPON | Inspiratory component IE ratio |
| E_IE_SPON | Expiratory component IE ratio |
| ELASTANCE_CMH2O_L | Elastance |
| RSB_S_L | Rapid shallow breathing index |
| COMP_DYN_MLS_CMH2O | Dynamic compliance |
| COMP_20_MLS_CMH2O | Compliance 20 |

TIME\_CONSTANT\_S Time constant

TIME\_CONSTANT\_EXPIRED\_S Time constant expired P01 CMH2O Airway occlusion pressure NIF CMH2O **Negative Inspiratory Force** EIP CMH2O **End inspiratory Pressure** 

FIO2 PC Fractional Inspired Oxygen VTCO2\_MLS Tidal CO2 production V\_CO2\_MLS\_MIN CO<sub>2</sub> Production

VOLUME\_DS\_MLS Deadspace Volume

ET\_CO2\_KPA End tidal CO2 kPa

ET\_CO2\_VOLPC End tidal CO2 vol% CO2\_SLOPE\_KPA\_L CO<sub>2</sub> Slope

Time low - Ventilator Setting

Maximum Inspiratory Time - Ver

Maximum time low - Ventilator :

Slope setting - Ventilator Setting

Partial Pressure CO2

| FLOW_SETTING_L_MIN | Flow setting - Ventilator Setting |
|------------------------------|------------------------------------|
| CONST_FLOW_L_MIN | Constant flow - Ventilator setting |
| RESPIRATORY_RATE_SETTING_MIN | Respiratory rate - Ventilator Sett |
| P_SUPPORT_SETTING_CMH2O | Pressure support - Ventilator Set |
| TIDAL_VOLUME_SETTING_MLS | Tidal volume setting - Ventilator |
| FLOW_TRIGGER_SETTING_L_MIN | Flow trigger - Ventilator Setting |
| ATC_COMPENSATION_SETTING_PC | ATC compensation - Ventilator S |
| FIO2_SETTING_PC | Fractional Inspired Oxygen - Ven |
| INSP_TERM_SETTING_PIF_PC | Inspiratory term % Peak Inspirat |
| EXP_TERM_SETTING_PIF_PC | Expiratory term % Peak Expirato |
| 11.1.4 Blood Gas Analysis | |
| STUDY_ID | Unique study data set identifier |
| DATETIME | ISO 8601 Date & Time |
| BLOOD_GAS_TYPE | Blood gas type |

T\_LOW\_SETTING\_S

SLOPE\_SETTING\_S

PCO2 KPA

T\_INSP\_MAX\_SETTING\_S

T\_LOW\_MAX\_SETTING\_S

| NA_MMOL_L | Sodium concentration |
|------------------------|--------------------------------|
| CL_MMOL_L | Chloride concentration |
| HAEMOGLOBIN_G_L | Haemoglobin concentration |
| OXY_HAEMOGLOBIN_PC | Oxyhaemoglobin |
| CARBOXY_HAEMOGLOBIN_PC | Carboxyhaemoglobin |
| H_HAEMOGLOBIN_PC | Deoxyhaemoglobin |
| METHE_HAEMOGLOBIN_PC | Methehaemoglobin |
| GLUCOSE_MMOL_L | Glucose concentration |
| LACTATE_MMOL_L | Lactate concentration |
| TEMP_BLOOD_GAS_C | Temperature blood gas |
| FIO2_BLOOD_GAS_F | FiO2 blood gas |
| R_BLOOD_GAS | Respiratory quotient |
| P50_BLOOD_GAS_KPA | P50 |
| BASE_EXCESS_MMOL_L | Base Excess |
| BASE_EXCESS_ACT_MMOL_L | Actual Base Excess |
| HCO3_MMOL_L | Bicarbonate concentration |
| HCO3_STAND_MMOL_L | Standardised bicarbonate conce |

# 11.1.1 ECMO

STUDY ID Unique study data set identifier

IN

| SWEEP_FO2_ECMO_ICIP_F | Sweep Gas Fractional O2 concer |
|----------------------------|----------------------------------|
| SWEEP_FLOW_ECMO_ICIP_L_MIN | Sweep gas flow |
| P_ACCESS_ECMO_CHELP_MMHG | Access pressure - Cardiohelp dat |
| P_PREOXY_ECMO_CHELP_MMHG | Pre membrane pressure - Cardio |
| P_POSTOXY_ECMO_CHELP_MMHG | Post membrane pressure - Cardi |
| P_TMP_ECMO_CHELP_MMHG | Transmembrane pressure - Card |
| Q_BLOOD_ECMO_CHELP_L_MIN | ECMO Blood Flow - Cardiohelp o |
| PUMP_ECMO_CHELP_RPM | ECMO Pump RPM - Cardiohelp d |
| SVO2_ECMO_CHELP_PC | Pre Membrane Haemoglobin sat |

## 11.2 Format and Scale of Data

The requirements and nature of this project mean that all study data will

Data will be collated to comma separated value (CSV) format. CSV is accessible by all major data processing software platforms e.g. spreads software. The vast majority of modern programming languages possess to format files.

The near universal interoperability of the CSV format ensures ease of data validity of collated data sets.

It is anticipated that this project will require several iterations of development, with each iteration examining a different treatment interviewill inform the exact nature of data collection in the subsequent iteration limited to the scope defined in the preceding section, 11.1

Collated data will then be subject to the defined anonymisation process, data will be made available to academic resorrepository.

## 11.4 Data Quality and Standards

Data retrieved from the EHR has been validated by a qualified clinician at be considered representative of patient condition and treatment.

Data retrieved from medical equipment, e.g. ventilators, is not validated data domains exhibit different qualities in this regard. Lab value measurements are made on equipment that is calibrated on a basis approhigh quality and safe care. Data from sources such as ventilators of standardised in that the equipment models are standardised across GSTF

## 11.5 Data handling and record keeping

The collaborative nature of this study requires that data be managed a environments:

- GSTFT
- Data Repository
- Academic partners

Please note the data pathway defined in section 7.2 of this document.

Each environment differs in available data management facilities a practices and compliance that must be observed. Each environment v separately.

#### 11.5.1 GSTFT

Data available at GSTFT can be of a personal and confidential nature, an project where the highest risk of breaching patient confidentiality exists.

N

- Confidentiality & Data Protection Policy (Version 2)
- Information Security Policy (Version 4)
- Information security (Principle f)

#### 11.5.2 Data Repository

This project will set up a central data repository for data storage and dist

Clinical investigators at GSTFT will upload data sets to the data repository. for ensuring the local and data repository indexes are maintained and up

GSTFT operates a SharePoint site, to which read only access can be given GSTFT.

The duplication between data sets stored within IT systems at GSTFT and as an extra layer of redundant storage and mutual back up.

Data storage, management and security practices for the data repository Operating Procedures (SOP):

 PSTOTICU\_SOP\_003 - Standard Operating Procedure Administrator

#### 11.5.3 Academic Partners

The University of Warwick (UWAR) and the University of Nottingham (UO of this study and are the end recipients of compiled data sets.

Data storage and management practices for study participants at UWA Standard Operating Procedure (SOP):

PSTOTICU\_SOP\_002 - Data Storage and Management by Ac

11 6 Metadata standards and data documentation

A log of study subjects linked to unique study data set identifiers investigators at GSTFT. This record will be securely stored within the site f form within GSTFT. This log will not be shared to the central repository oblank log is provided by study document:

PSTOTICU SD 004 – Subject Log

A full index of the collated subject data set files will be maintained by silocal GSTFT copy will be kept, and duplicated within the central data repeindex is included in ****, and a blandocument:

PSTOTICU SD 005 – Data Set Index

## 11.6.2 Metadata Descriptive Files

provide a more accessible context for the data.

To provide context for the CSV files of a data set, text files will be a describing the intervention captured. These descriptions will be entirely lintervention and provide no data which might provide an increased subjects. File format will be of a txt format, and thus universally readable textual descriptions will be apparent on examination of the quantitative

#### Example descriptions:

- 'PEEP increased from 5cmH2O to 10cmH2O'
- '250ml Crystalloid Bolus given at 02:00' \*
  - 'Prone positioning started 02:00. Prone positioning disc
- \* Dates and times are subject to anonymisation as per PSTOTICU\_SO Procedure (SOP) Data De-Identification

#### 11.7 Data preservation strategy and standards

The data repository will be maintained for a five year period after da completed. After this period, access will be revoked for those users with will be retained as part of the study archival process at GSTFT and duplicano longer required.

#### 11.7.3 Academic Collaborators

Upon completion of data collection activities, it is anticipated that acade extended period. Data will be available to project collaborators for five activities are completed.

# 11.8 Data Security and Confidentiality of Potentially Information

The level of data security is dependent upon the nature of the data – per higher levels of security.

Data collected for this study will be subjected to an anonymisation proce a negligible risk of subject re-identification.

Despite the low risk of subject identification, health related data is appropriate to ensure study data is handled in a way that ensures sagainst unlawful or unauthorised processing, access, loss, destruction or

## 11.8.1 Data Anonymisation

The aim of anonymisation, is to ensure that the risk of potential re-iden minimised to negligible levels.

Clinical data will be collected by investigators at GSTFT and subject anonymisation process, before being made available to academic partners anonymisation process employed is defined in the SOP:

PSTOTICU SOP 004 – Standard Operating Procedure (

Data will be stored on GSTFT network drives within a proje S:\IntensiveCare\Research folder. This ensures that access to data is Intensive Care clinical research team at GSTFT. Access is authoris authorisation system administered by GSTFT IT services and therefore to the security of clinical services and data. This method of project specificacross the research portfolio of this research team.

Usage of GSTFT network drives also ensures the durability and availability same standard as that provided for clinical services and data.

GSTFT data management practice and information governance policy will is resident within the GSTFT environment.

## 11.8.2.2 Data Repository

Access to the data repository requires a username and password, and ex an additional one time pass code is required. One time pass codes are authentication app set up at the time of account registration.

Authorisation and permissions are described in the Standard Operating F

 PSTOTICU\_SOP\_003 - Standard Operating Procedure Administrator

The clinical investigator team at GSTFT will have permissions to upload and collaborators will be granted read only permissions to the repository, a download data sets and indexes only.

Auditing of all file operations and specifically downloads will be implementable trail of repository activity is available. This will be collated, reviewed and monthly basis.

Data sets stored in the repository will be duplicates of data stored within

N

Data will only be processed on specific computing devices maintained with Storage on project computers will be encrypted with BitLocker software a over an encrypted transport layer. Access to project computers will be lin

Potential loss of data from the computing environments of study collaboration of data within the repository and GSTFT environments.

## 11.9 Data Collection and Processing Responsibilities

The chief investigator for this project has ultimate responsibility for engadministered in accordance with the processes outlined by this SOP.

The chief investigator may delegate responsibility for management of the clinical investigators. A record of delegated responsibilities will be maintaged the study document:

PSTOTICU\_SD\_008 – Staff Delegation Log

## 12 Statistical considerations

#### 12.1 Sample size calculation

The subjects will comprise a convenience sample only. This study is not size or incidence, and so a formal sample size calculation to ensure inappropriate. Power calculation is not meaningful in this context, si prospective matching technology rather than statistical comparison.

As described in section 8, the admission of one patient may contribute catalogue of data sets within the repository.

The iterative nature of model development was described previously in so that there will a large but variable number of episodes, fitting the require iteration, available from the electronic health record.

Although the precise number of iterations or available episodes cannot anticipate 20 development iterations for which a maximum of 250 approve thus put an upper bound of collected episodes at 5,000 episodes.

# 12.2 Statistical analysis

vasoconstriction.

The core models have been designed to represent a dynamic in vivo card

The pulmonary model is comprised of conducting airways and a resp alveolar compartments, with each compartment having a corresponding s for stiffness, threshold opening pressures and extrinsic pressures as wel vascular resistances. This allows for a wide spectrum of ventilation replicated. The model includes inherent physiological reflex mechanis

The cardiovascular model consists of 19 vascular compartments, each momentary pressure and volume and its non-linear compliance. Ventricularing a time-dependent elastance, which implements pulsatile blood flo

is variably transmitted to all intrathoracic compartments, including the

## 13 Ethical considerations

HRA approval will be sought for this study. Local R&D approval will also be

# 14 Financing and Insurance

Finance for this project is provided through an EPSRC grant, reference nu

Insurance is provided by the sponsor, Guys & St Thomas' NHS Foundation

# 15 Reporting and dissemination

Progress of the study will be disseminated and discussed at collaborator

The findings will be presented at national and international conferences a journals.

- Chikhani, M., Das, A., Haque, M., Wang, W., Bates, D., & Hardman, J. respiratory distress syndrome: quantutative evaluation be oxygenation and decreased oxygen delivery. *British Journal of Ar*
- Das, A., Cole, O., Chikhani, M., Wang, W., Ali, T., Haque, M., . . . Hardman recruitment maneuvers in acute respiratory distress. *Critical Care*
- Das, A., Haque, M., Chikhani, M., Cole, O., Wang, W., Hardman, J., & Bate effects of lung recruitment maneuvers in acute respirator distress *Medicine*, *17*, 34.
- Hardman, J., Bedforth, N., Ahmed, A., Mahajan, R., & Aitkenhead, A. (19 validation of its respiratory components and its ability to predict changes in mechanical ventilation. *British Journal of Anaesthesia*.
- Laviola, M., Das, A., Chikhani, M., Bates, D., & Hardman, J. (2017). Investoscillations and deadspace gas mixing during apnea using complete Eng Med Biol Soc, 337-340.
- Laviola, M., Das, A., Chikhani, M., Bates, D., & Hardman, J. (2019). Comechanisms of carbon dioxide clearance. *British Journal of Anaes*
- McCahon, R., Columb, M., Mahajan, R., & Hardman, J. (2008). Validation fidelity, computational model of acute respiratory distress synd the indices of oxygenation at constant lung-state. *British Journal* 365.
- McNamara, M., & Hardman, J. (2005). Hypoxaemia during open-airwa modelling analysis. *Anaesthesia*, *60*, 741–746.